CLINICAL TRIAL: NCT01798745
Title: A Randomized, Double-blind, Placebo-controlled Pharmacokinetic and Pharmacodynamic Two Part Cohort Study of JNJ-54452840 in Subjects With Reduced Systolic Function Heart Failure and Elevated Levels of Anti-Beta 1 Adrenergic Receptor Autoantibodies
Brief Title: A Study to Assess the Pharmacokinetics and Pharmacodynamics of JNJ-54452840 in Participants With Heart Failure and Anti-beta1-adrenergic Receptor Autoantibodies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study not required for development
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100985; 54452840HFA2003 (Other: Janssen Research & Development LLC); 2012-005302-22 (EudraCT Number)
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Heart Failure
Keywords: Heart failure; JNJ-54452840; Anti-beta-1 adrenergic receptor auto antibodies; Beta-1 adrenergic receptor; Antibodies; Auto antibodies; Systolic function
MeSH Terms: conditions — Heart Failure | interventions — JNJ-54452840

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Cohort A: JNJ-54452840 20 mg (Experimental): Each patient will receive 20 mg of JNJ-54452840 as a single dose.
  Interventions: Drug: JNJ-54452840
- Cohort A: JNJ-54452840 80 mg (Experimental): Each patient will receive 80 mg of JNJ-54452840 as a single dose.
  Interventions: Drug: JNJ-54452840
- Cohort A: JNJ-54452840 160 mg (Experimental): Each patient will receive 160 mg of JNJ-54452840 as a single dose.
  Interventions: Drug: JNJ-54452840
- Cohort A: Placebo (Placebo Comparator): Each patient will receive matching placebo as a single dose.
  Interventions: Other: Placebo
- Cohort B: JNJ-54452840 <= 240 mg (Experimental): Each patient will receive JNJ-54452840 at a dose of less than or equal to 240 mg as a single dose (dose determined by the Data Monitoring Committee).
  Interventions: Drug: JNJ-54452840
- Cohort B: Placebo (Placebo Comparator): Each patient will receive matching placebo as a single dose.
  Interventions: Other: Placebo
- Cohort C: JNJ-54452840 for 3 days (Experimental): Each patient will receive JNJ-54452840 once daily for 3 days at a dose determined by the Data Monitoring Committee (daily dose not exceeding 240 mg).
  Interventions: Drug: JNJ-54452840
- Cohort C: Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 3 days.
  Interventions: Other: Placebo
- Cohort D: JNJ-54452840 for 5 days (Experimental): Each patient will receive JNJ-54452840 once daily for 5 days at a dose determined by the Data Monitoring Committee (daily dose not exceeding 240 mg).
  Interventions: Drug: JNJ-54452840
- Cohort D: Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 5 days.
  Interventions: Other: Placebo
- Cohort E: JNJ-54452840 weekly (Experimental): Each patient will receive JNJ-54452840 once weekly on Days 1, 8, 15, and 22 at a dose determined by the Data Monitoring Committee (daily dose not exceeding 240 mg).
  Interventions: Drug: JNJ-54452840
- Cohort E: Placebo (Placebo Comparator): Each patient will receive matching placebo once weekly on Days 1, 8, 15, and 22.
  Interventions: Other: Placebo
- Cohort F: JNJ-54452840 multiple dose (Experimental): Each patient will receive JNJ-54452840 once daily (for 3 or 5 days) or once weekly (up to Day 22) as determined by the Data Monitoring Committee and as explored in Cohorts C, D, and E (daily dose not exceeding 240 mg).
  Interventions: Drug: JNJ-54452840
- Cohort F: Placebo (Placebo Comparator): Each patient will receive matching placebo once daily (for 3 or 5 days) or once weekly (up to Day 22).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JNJ-54452840 — Once daily intravenous injection(s) (medication is injected into a vein) at doses ranging from 20 mg to 240 mg, given as a single injection (Cohorts A and B); injections given once daily over 3 to 5 days (Cohorts C, D, and F); or injections given once weekly up to Day 22 (Cohorts E and F).
  Arms: Cohort A: JNJ-54452840 160 mg; Cohort A: JNJ-54452840 20 mg; Cohort A: JNJ-54452840 80 mg; Cohort B: JNJ-54452840 <= 240 mg; Cohort C: JNJ-54452840 for 3 days; Cohort D: JNJ-54452840 for 5 days; Cohort E: JNJ-54452840 weekly; Cohort F: JNJ-54452840 multiple dose
Other: Placebo — Once daily matching intravenous injection(s) (medication is injected into a vein) given as a single injection (Cohorts A and B); injections given once daily over 3 to 5 days (Cohorts C, D, and F); or injections given once weekly up to Day 22 (Cohorts E and F).
  Arms: Cohort A: Placebo; Cohort B: Placebo; Cohort C: Placebo; Cohort D: Placebo; Cohort E: Placebo; Cohort F: Placebo

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of JNJ-54452840 in participants with heart failure and anti-beta1-adrenergic receptor autoantibodies. The safety and tolerability of JNJ-54452840 will also be assessed.

DETAILED DESCRIPTION:
This study will be randomized (the study treatment is assigned by chance), double-blind (neither investigator nor participant knows the treatment received), and placebo-controlled (one of the study treatments is inactive). This study will be conducted in participants with reduced systolic function heart failure (a reduced amount of blood is pumped around the body compared with a normal heart) and elevated levels of anti-beta1-adrenergic receptor autoantibodies (antibodies that may be involved in development, progression, or worsening of heart failure). The study will be conducted in 2 parts; participants will receive single doses of JNJ-54452840 in Part 1 and multiple doses in Part 2. Each part of the study will consist of 3 phases; a screening phase, a double-blind treatment phase, and a follow-up phase. There will be 2 cohorts (groups) of participants in Part 1 of the study. In Part 1 (Cohort A), participants will be randomly assigned to 1 of 4 treatment groups: a single intravenous (medication is injected into a vein) dose of 20 mg JNJ-54452840; a single intravenous dose of 80 mg JNJ-54452840; a single intravenous dose of 160 mg JNJ-54452840; or matching placebo (inactive medication). In Part 1 (Cohort B), participants will be randomly assigned to 1 of 2 treatment groups; a single intravenous dose of less than or equal to 240 mg JNJ-54452840 (as determined by the Data Review Committee after review of Cohort A data) or matching placebo. There will be 4 cohorts of participants in Part 2 of the study; the dose of JNJ-54452840 used in each cohort, initiation of each cohort, and the sequence will be decided by the Data Review Committee. In Part 2 (Cohort C), participants will be randomly assigned to 1 of 2 treatment groups: JNJ-54452840 or matching placebo given intravenously once daily for 3 days. In Part 2 (Cohort D), participants will be randomly assigned to 1 of 2 treatment groups: JNJ-54452840 or matching placebo given intravenously once daily for 5 days. In Part 2 (Cohort E), participants will be randomly assigned to 1 of 2 treatment groups: JNJ-54452840 or matching placebo given intravenously once weekly on Days 1, 8, 15, and 22. In Part 2 (Cohort F), participants will be randomly assigned to 1 or more treatment groups involving regimen(s) as explored in Cohorts C, D, or E. Single doses of JNJ-54452840 will not be greater than 240 mg for any Cohort. The active to placebo randomization ratio for each cohort following Cohort A (ie, Cohorts B, C, D, E, and F) will be determined by the Data Review Committee. Participants will come to the study center each time they receive study medication and will remain at the center for at least two hours following each injection. Blood samples will be drawn at time points during the screening period and treatment period for participants in both Part 1 and Part 2 of the study. Participants will return to the study center after the double-blind treatment phase on Day 29 and then for follow-up visits on Days 57 and 85. Participants in Part 1 or Part 2 will be involved in the study for approximately 112 days. Participant safety will be monitored. The study drug, JNJ-54452480 is being investigated for the treatment of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented medical history of symptomatic (ie, showing symptoms) reduced ejection fraction (measurement of the percentage of blood leaving the heart each time it contracts) heart failure due to either ischemic etiology (decreased blood supply to heart) or non-ischemic dilated cardiomyopathy (heart is weakened and enlarged) for at least 4 months prior to the screening visit
* Must have heart failure classified by the New York Heart Association classification system as class I through IIIa
* Must have a left ventricular ejection fraction (measurement of the percentage of blood leaving the heart each time it contracts) of < = 45%
* Must have blood levels of anti-beta1-adrenergic receptor autoantibodies (antibodies that are involved in developing heart failure) that are above the reference range
* Must have been receiving guideline-directed medical therapy for heart failure for at least 4 months prior to screening and, in addition, be receiving stable and individually optimized drug doses for at least 2 months prior to screening.

Exclusion Criteria:

* History of, or current active illness that, in the opinion of the investigator, would make participation not in the best interest (eg, compromise the well-being) of the patient or that could interfere with the study assessments
* Left ventricular end-diastolic diameter index (a measure of the heart's performance) of <= 32 mm/m2
* N-terminal pro-brain natriuretic peptide level (a biologic molecule that has been shown to predict cardiac events) that is <= 200 pg/mL in participants with normal sinus rhythm or <= 800 pg/mL in participants with atrial fibrillation
* Chronic treatment with immunosuppressive drugs (except for <= 5 mg/day prednisone-equivalent dose)
* Known allergies to peptides or proteins, such as albumin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serum levels of anti-beta1-adrenergic receptor autoantibody bound JNJ-54452840 | Up to Day 7
  Serum levels of bound JNJ-54452840 (ie, amount of drug that is attached to anti-beta1-adrenergic receptor autoantibodies) will be used to determine pharmacokinetic parameters for JNJ-54452840 (measurements describing how the body affects the drug).
Serum levels of free JNJ-54452840 | Up to Day 7
  Serum levels of free JNJ-54452840 (ie, amount of drug that is not attached to anti-beta1-adrenergic receptor autoantibodies) will be used to determine pharmacokinetic parameters for JNJ-54452840 (measurements describing how the body affects the drug).
Serum levels of total JNJ-54452840 | Up to Day 7
  Serum levels of total JNJ-54452840 (ie, bound drug plus free drug) will be used to determine pharmacokinetic parameters for JNJ-54452840 (measurements describing how the body affects the drug).
Serum levels of anti-beta1-adrenergic receptor autoantibodies | Up to Day 85
  Blood levels of anti-beta1-adrenergic receptor autoantibodies will be used to determine the pharmacodynamics of JNJ-54452840 (ie, how the drug affects the body).
Beta1-adrenergic receptor activation | Up to Day 29
  Beta1-adrenergic receptor activation will be used to determine the pharmacodynamics of JNJ-54452840 (ie, how the drug affects the body).

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to Day 85
  Number of patients with adverse events will be used as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.